CLINICAL TRIAL: NCT05320718
Title: Comparison of Programmed Intermittent Bolus Infusions of Spinae Plane Block Versus Paravertebral Block for Analgesia in Minimally Invasive Direct Coronary Artery Bypass Grafting
Brief Title: Analgesia in Minimally Invasive Direct Coronary Artery Bypass Grafting: Programmed Intermittent Bolus Infusions of Erector Spinae Plane Block Versus Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Principal Investigator, Min Li, Vice Director of the Department of Anesthesiology, Principal Investigator, Clinical Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESPB vs PVB for MIDCAB
Record Dates: First submitted 2022-03-21; First posted 2022-04-11 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Regional Anesthesia; Anesthesia, Local; Surgery
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- erector spinae plane block (Experimental): A needle is inserted until the tip contacted the T5 transverse process under ultrasound guidance. After confirming the needle tip position, 20 ml of 0.5% ropivacaine was injected in the plane between the erector spinae muscles and transverse process. A catheter is inserted through the needle and then connected to a Programmed Electronic Postoperative Analgesia Pump with a programmed intermittent bolus of 10 ml ropivacaine 0.2% every 2 h after surgery
  Interventions: Drug: Ropivacaine
- thoracic paravertebral block (Active Comparator): A needle is inserted into the paravertebral space. After confirming the needle tip position, 20 ml of 0.5% ropivacaine is injected in the paravertebral space. A catheter is inserted through the needle and then connected to a Programmed Electronic Postoperative Analgesia Pump with a programmed intermittent bolus of 10 ml ropivacaine 0.2% every 2 h after surgery.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 20 ml of 0.5% ropivacaine as bolus and a programmed intermittent bolus of 10 ml ropivacaine 0.2% every 2 h after surgery

SUMMARY:
Paravertebral block (PVB) has been regarded as effective regimen for pain control after cardiac surgery. As a novel analgesia technique, erector spinae plane block (ESPB) has been reported to provide effective analgesia after thoracic and cardiac surgery. We hypothesized that the ESPB is non-inferior to PVB in treating pain in minimally invasive direct coronary artery bypass surgery.

DETAILED DESCRIPTION:
Minimally invasive direct coronary artery bypass grafting has recently gained with popularity in treatment of coronary artery disease. Compared with conventional approach, it has advantages of less trauma and rapid recovery, but postoperative pain is severe, which may increase the risk of cardiopulmonary complications and cause chronic pain. Therefore, perioperative analgesia is crucial in minimally invasive direct coronary artery bypass grafting.

Paravertebral block (PVB) has been regarded as effective regimen for pain control after cardiac surgery. As a novel analgesia technique, erector spinae plane block (ESPB) has been reported to provide effective analgesia after thoracic and cardiac surgery. We hypothesized that the ESPB is non-inferior to PVB in treating pain in minimally invasive direct coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective minimally invasive direct coronary artery bypass grafting

Exclusion Criteria:

1. Contraindications to regional anesthesia (coagulopathy, infection of the skin at the site of needle puncture area, et al)
2. Morbid obesity (body mass index > 35 kg/m2)
3. Allergy to any of the study drugs
4. Chronic opioid use or history of opioid abuse.
5. Inability to understand pain score

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
pain at cough after surgery | postoperatively 0-3 day
  Numerical Rating Pain Scale, where 0=No Pain (better outcome) and 10=Intractable Pain (worse outcome)
postoperative rescue analgesic consumption | postoperatively 0-3 day
  morphine equivalents

SECONDARY OUTCOMES:
pain at rest after surgery | postoperatively 0-3 day
  Numerical Rating Pain Scale, where 0=No Pain (better outcome) and 10=Intractable Pain (worse outcome)
adverse events of regional block | Intraoperative (during and immediately after block performance)
  local bleeding, pleural puncture, local anesthetic toxicity
dermatome of block | immediately after extubation
  loss of cold sensation (ice cubes), 3-point scale: 0 = loss of cold sensation, 1=decreased cold sensation, 2 = normal sensation.

OTHER OUTCOMES:
pulmonary function | preoperative and postoperative day 1 and 3
  parameters measured by bedside spirometer, FVC, FEV1, FEV1/VC, FEF25%, FEF50%, FEF25-75, PEF
postoperative complications: cardiac, pulmonary, cerebral, opioid intake | 3 days postoperatively
  incidence of severe arrhythmia, cardiac arrest, pneumonia, atelectasis, pulmonary edema, postoperative delirium, nausea, vomiting
recovery time | postoperatively, up to 4 weeks
  Time for extubation, oral intake, chest drain tube removal, discharge from ICU and discharge from hospital
plasma cortisol | preoperative, 24 hours and 72 hours after operation.
  The investigator will measure the plasma cortisol level at several time points
C-reactive protein | preoperative, 24 hours and 72 hours after operation.
  The investigator will measure the plasma C-reactive protein level at several time points
plasma troponin T level | preoperative, 24 hours and 72 hours after operation.
  The investigator will measure the plasma troponin T level at several time points
patient's satisfaction with regional analgesia | 3 day postoperatively
  Patient overall satisfaction with regional analgesia will be assessed on a 11 point scale, 0=not satisfied at all, 10=extremely satisfied
time to perform the block | immediately before surgery
  from identify the landmark using ultrasound to catheter fixation
CK-MB | preoperative, 24 hours and 72 hours after operation
  The investigator will measure the plasma CK-MB level at several time points
performance in activities of daily living (ADL) | 3 month and 6 month postoperatively
  Post-operative follow-up phone calls will be used to assess performance in activities of daily living (ADL) with the Barthelindex of ADL

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, MD, Principal Investigator — Peking University Third Hospital
Locations (2):
- China (2):
  - Department of Anesthesiology,Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University Third Hosptial, Beijing

REFERENCES:
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH. Erector spinae plane block and thoracic paravertebral block for breast surgery compared to IV-morphine: A randomized controlled trial. J Clin Anesth. 2020 Feb;59:84-88. doi: 10.1016/j.jclinane.2019.06.036. Epub 2019 Jul 4. PMID 31280100
- [Background] Saadawi M, Layera S, Aliste J, Bravo D, Leurcharusmee P, Tran Q. Erector spinae plane block: A narrative review with systematic analysis of the evidence pertaining to clinical indications and alternative truncal blocks. J Clin Anesth. 2021 Feb;68:110063. doi: 10.1016/j.jclinane.2020.110063. Epub 2020 Oct 5. PMID 33032124
- [Background] Huang W, Wang W, Xie W, Chen Z, Liu Y. Erector spinae plane block for postoperative analgesia in breast and thoracic surgery: A systematic review and meta-analysis. J Clin Anesth. 2020 Nov;66:109900. doi: 10.1016/j.jclinane.2020.109900. Epub 2020 Jun 2. PMID 32502778